CLINICAL TRIAL: NCT05110378
Title: Do Good Non-Technical Skills Correlate With Good Clinical Outcomes in Endoscopy?
Status: Completed | Type: Observational
Sponsor: University Hospital Plymouth NHS Trust (Other)
Collaborators: Torbay and South Devon NHS Foundation Trust (Other); Plymouth University Peninsula Schools of Medicine & Dentistry (Unknown)
Responsible Party: Sponsor
Other Study IDs: 15/P/101
Record Dates: First submitted 2018-12-18; First posted 2021-11-05 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Bowel Cancer
Keywords: non-technical skills; gastrointestinal endoscopy; qualitative research; training; assessment
MeSH Terms: conditions — Intestinal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Failures in non-technical skills (NTS) contribute to adverse events in healthcare. Previous research has explored the assessment and training of these skills, and yet there is a lack of evidence for their impact on clinical outcomes. Gastrointestinal endoscopy is a high-pressure specialty, but to date there is little on the role of NTS in this area, or a method for their assessment.

This MD project aims to measure NTS in endoscopy, explore their relationship with clinical outcomes, and identify those specific to this area of healthcare.

Methods An observational study of endoscopy teams in real time, using the Oxford NOTECHS II assessment tool. Comparison of NTS performance with procedure outcomes and patient satisfaction.

A qualitative interview study with staff members to establish the NTS specifically relevant to working in gastrointestinal endoscopy.

DETAILED DESCRIPTION:
Ten to fifteen percent of patients will experience some kind of adverse event during their hospital stay. A significant proportion of these occur in surgery. The causes of such adverse events often stem not from deficiencies in clinical or technical skills but from the non-technical aspects of human and team performance).

Much of the early research in this field comes from the aviation industry where "non-technical skills" are defined as "the cognitive and social skills of flight crew members in the cockpit". Failures in teamwork in cockpit crews have been linked to half of adverse events in aviation and further work within surgery has shown a significant reduction in adverse events when teams perform well.

Behavioural ratings systems have been used in aviation and other high risk industries for many years to facilitate assessment and training. "NOTECHS" was designed in the 1990s by a collaboration of European aviation experts as a system to assess the non-technical skills of individual pilots. Over recent years similar such tools or taxonomies have been developed in healthcare. Within surgery some taxonomies assess individual team members such as 'Non-Technical Skills for Surgeons' (NOTSS), 'Anaesthetists' Non-Technical Skills' (ANTS) and 'Scrub Practitioners List of Intra-operative Non-Technical Skills' (SPLINTS), whilst others aim to assess the whole team: 'revised NOTECHS', 'Oxford NOTECHS (II)' and 'Observational Teamwork Assessment for Surgery' (OTAS). 'NOTSS', 'ANTS' and 'SPLINTS' were developed by a group at the University of Aberdeen. Each provides a rating scale to assess the non-technical skills of an individual practitioner within a surgical team. They can be used as an observational assessment or a self-evaluation tool for reflection and professional development. The "revised NOTECHS" scale developed by a team at Imperial College, adapted the "NOTECHS" system to assess the non-technical skills of theatre teams. The "Oxford NOTECHS" was similarly adapted from "NOTECHS" to assess theatre teams but with an additional subdivision into three "sub-teams" (surgical, anaesthetic and nursing). The "Oxford NOTECHS" has further been revised to the "Oxford NOTECHS II" scale to improve the discrimination between levels of performance. "OTAS" combines a task checklist and a team behaviour assessment in the pre- operative, operative and post-operative phases of a procedure.

Two studies using the Oxford NOTECHS system have shown an improvement in scores after a training intervention. Mishra et al observed 65 laparoscopic cholecystectomies before and after a Crew Resource Management (CRM) style training intervention applied to all staff members (29 laparoscopic cholecystectomies before, 39 after). Oxford NOTECHS scores improved significantly after the training intervention. Scores negatively correlated with technical error rates and positively (but not significantly) with staff safety attitudes. Another study observing laparoscopic cholecystectomy and carotid endarterectomy showed similar improvement in Oxford NOTECHS scores after a training intervention (all staff trained). This was associated with a concurrent decrease in technical errors, procedural errors and an increase in Safety Attitude Questionnaire scores, but no significant change in clinical outcomes. These findings are consistent with a number of other studies investigating the effect of human factors team training within healthcare. Outcome measures vary between studies: learning assessment questionnaires, observed teamwork behaviour, participant perception of teamwork and staff attitudes have all been used as markers of performance and have all shown to improve after team training interventions. Unfortunately only a few studies have linked training interventions to clinical outcome improvements. The Veterans Health Administration Medical Team Training (MTT) program was a multi-center quality improvement program in the USA. This study showed a significant reduction in surgical morbidity after the introduction of team training. This along with the Oxford NOTECHS studies demonstrates that improving non-technical skills may improve clinical outcomes. Thus though there is a range of data on the effect of training on reduction of non-technical error, and some data which demonstrates a direct link between non-technical skills and successful outcomes, there is still much work to be done in clarifying the three-way links between non-technical skills, successful outcomes and the role of training.

Endoscopy units are akin to day-case theatre complexes. Endoscopic procedures vary in their length and complexity. Diagnostic gastroscopy and colonoscopy with or without biopsy (removal of tissue) are the commonest procedures performed. However, there are a wide range of therapeutic procedures also undertaken including stenting, endoscopic resection of tumours, endoscopic retrograde cholangio-pancreatography and feeding gastrostomy insertion. Patients consent to undergo these procedures having been fully informed of the risks involved. They are either awake, under sedation (56.4% of sedation in the Peninsula region occurs in Endoscopy units), or under general anaesthetic depending on the complexity of the procedure and their preference. The PHNT endoscopy unit performs more than 12,000 procedures per year in a contained unit of 5 rooms, operating Monday to Saturday. Additional procedures requiring x-ray screening occur within the radiology department supplemented by Endoscopists and Nursing staff from the unit.

There are clear auditable outcome standards for technical performance and training in Endoscopy provided by the British Society of Gastroenterology (BSG) and the Joint Advisory Group on GI Endoscopy (JAG). These include markers of completion of procedures such as Caecal Intubation Rate and Adenoma Detection Rate in Colonoscopy. Challand et al showed that good clinical performance in Colonoscopy was associated with increased efficiency. They also found that there was no negative effect of training on either of these outcomes.

Although adverse events are rare in Endoscopy, advances in technology and techniques have led to an increase in risk. As therapeutic procedures become more advanced the more "surgical" the specialty becomes. The National Confidential Enquiry into patient Outcomes and Death Report 2004 investigated the death of 1818 patients within 30 days of therapeutic endoscopy during April 2002 to March 2003. They found a wide variety of practice in different units across the UK, particularly in areas such as sedation administration, patient monitoring and planning of procedures: the non-technical aspects of endoscopy.

The Endoscopist, whether a Surgeon, Physician or Advanced Nurse Practitioner, is equivalent to the operating surgeon and nursing staff perform very similar roles to theatre nurses/practitioners. An anaesthetist is present only for those procedures performed under general anaesthetic. Despite a similar team and technical set up to an operation room there is a clear deficit in the literature with regards to non-technical skills and team performance within Endoscopy. It is likely that there will be a three-way relationship between non-technical skills, successful outcomes and training as there are for other surgical areas.

Endoscopy units share many characteristics with theatre complexes and are pioneering increasingly complex procedures and yet there is little literature relating to the assessment or training of team performance in this area; even within other areas of healthcare there is little correlation with clinical outcomes. Taxonomies for team performance and non-technical skills assessment in surgery are now well established and yet there still is no published evidence of their use in or adaptation for Endoscopy. There is therefore scope for:

1. The evaluation and development of a non-technical skills assessment tool within Endoscopy (based on Oxford NOTECHS II - a well-established taxonomy with good reliability and validity). Correlation of non-technical skills with clinical and other outcomes. Our endoscopy unit has a large throughput of similar cases per annum (>12,000). This means the face, construct and concurrent validity of the non-technical skills assessment tool can be tested reliably with greater power. Scores could be correlated easily with standardized quality and safety outcomes.
2. Development of a Human Factors Simulation team training intervention based on the knowledge gained from. Training has yet to take place within the Endoscopy unit in our Hospital.

The aims of the project are as follows:

To develop the measurement of non-technical skills in endoscopy (using the Oxford NOTECHS II taxonomy); to delineate the relationship between successful clinical (and other) outcomes and non-technical skills as measured by the tool.

Endoscopy units share many characteristics with theatre complexes and are pioneering increasingly complex procedures and yet there is little literature relating to the assessment or training of team performance in this area; even within other areas of healthcare there is little correlation with clinical outcomes. Taxonomies for team performance and non-technical skills assessment in surgery are now well established and yet there still is little evidence of their use in or adaptation for Endoscopy. This project seeks to provide a firm basis for future work by establishing the measurement of non-technical skills in endoscopy, relating those skills to clinical outcomes, and identifying those features of non-technical skills training likely to be of greatest importance in terms of successful clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

Staff

* Endoscopy staff consenting to take part in the study
* Staff work in Endoscopy as their main NHS job Patients
* Patients consenting to be observed and complete a patient satisfaction survey
* Male or Female, aged 18 years or above
* Able (in the investigator's opinion) and wiling to comply with all study requirements

Exclusion Criteria:

Staff • Endoscopy staff not consenting to take part in the study

Patients

* Patients not consenting to take part in the study
* Patients unable to understand the information provided or give consent to participate

  o This was determined by the researcher who in her role as surgical doctor has been trained to assess patients' capacity to give informed consent.
* Aged less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Endoscopy staff (medical and non-medical) at Plymouth Hospitals NHS Trust and Torbay and South Devon NHS Foundation Trust.
  Patients attending the Endoscopy department during the study period were provided with written information explaining the study and inviting them to take part.
Sampling Method: Non-Probability Sample
Enrollment: 326 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-10-04 (Actual); Study Completion 2018-01-24 (Actual)

PRIMARY OUTCOMES:
Oxford NOTECHS II | 100 endoscopic procedures over a period of 4-5 weeks
  A Modified Theatre Team Non-Technical Skills Scoring System

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Ward, BSc, MBBS, FRCA, PGCME, Study Chair — University Hospitals Plymouth NHS Trust; Charlotte Hitchins, BMedSci, BMBS, MRCS, Principal Investigator — University Hospitals Plymouth NHS Trust

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hitchins CR, Metzner M, Edworthy J, Ward C. Non-technical skills and gastrointestinal endoscopy: a review of the literature. Frontline Gastroenterol. 2018 Apr;9(2):129-134. doi: 10.1136/flgastro-2016-100800. Epub 2017 Mar 29. PMID 29588841